CLINICAL TRIAL: NCT00571519
Title: A Randomized, Double-blind, Placebo, and Active Comparator-controlled, Parallel-group Study of the Efficacy and Safety of Rivoglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Brief Title: Randomized, Double-blind, Active-controlled, Study of Rivoglitazone in Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSPD focusing on Study 301 to confirm the clinical profile before proceeding. Daiichi Sankyo Pharma Development terminated this study on 23 Apr 2008 because of changes in the clinical development plan with 94 of 2600 planned, randomized participants.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS0011-A-U302
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- 1 (Experimental): rivoglitazone HCl 0.5mg
  Interventions: Drug: Rivoglitazone HCl; Drug: metformin
- 2 (Experimental): rivoglitazone HCl 1.0 mg
  Interventions: Drug: rivoglitazone HCl; Drug: metformin
- 3 (Experimental): rivoglitazone HCl 1.5 mg
  Interventions: Drug: rivoglitazone HCl; Drug: metformin
- 4 (Placebo Comparator): placebo matching rivoglitazone HCl tablets
  Interventions: Drug: placebo; Drug: metformin
- 5 (Active Comparator): pioglitazone HCl 15 mg
  Interventions: Drug: pioglitazone HCl; Drug: metformin
- 6 (Active Comparator): pioglitazone HCl 30 mg
  Interventions: Drug: pioglitazone HCl; Drug: metformin
- 7 (Active Comparator): pioglitazone HCl 45 mg
  Interventions: Drug: pioglitazone HCl 45 mg; Drug: metformin
- 8 (Placebo Comparator): matching placebo for pioglitazone
  Interventions: Drug: placebo; Drug: metformin

INTERVENTIONS:
Drug: Rivoglitazone HCl — 0.5 mg tablets administered orally, once daily
  Other Names: CS-011
  Arms: 1
Drug: rivoglitazone HCl — 1.0 mg tablets administered orally, once daily
  Other Names: CS-011
  Arms: 2
Drug: rivoglitazone HCl — 1.5 mg tablets administered orally, once daily
  Other Names: CS-011
  Arms: 3
Drug: placebo — placebo tablets matching rivoglitazone tablets administered orally, once daily
  Arms: 4
Drug: pioglitazone HCl — 15 mg capsules administered orally, once daily
  Arms: 5
Drug: pioglitazone HCl — 30 mg capsules administered orally, once daily
  Arms: 6
Drug: pioglitazone HCl 45 mg — 45 mg capsules administered orally, once daily
  Arms: 7
Drug: placebo — placebo capsules for pioglitazone administered orally, once daily
  Arms: 8
Drug: metformin — Oral tablets. Rescue medication.

SUMMARY:
This is a 26-week, multicenter, randomized, double-blind, placebo and active comparator-controlled, parallel-group study in participants with type 2 diabetes currently sub-optimally controlled by diet and exercise or with non-thiazolidinedione antihyperglycemic monotherapy. Pioglitazone is used as active comparator. The total duration of a participant's participation will be approximately 30 weeks, including a 2-week placebo lead-in period, a 26-week double-blind treatment period, and a 2-week post-treatment follow-up period. Participants who complete the randomized portion of the study per protocol may have the opportunity to continue in a long-term extension study of active treatments.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent at screening.
* Diagnosed with type 2 diabetes mellitus.
* Glycosylated hemoglobin (A1c) >7.0% and ≤8.5% at screening.
* Male or female ≥18 years of age.
* Women of childbearing potential must have been using an adequate method of contraception to avoid pregnancy throughout the study, and for up to 4 weeks after study completion.
* Fasting C-peptide level >0.5 ng/mL at screening.
* Currently being treated with a stable dose of an approved non-thiazolidinedione antihyperglycemic medication (including sulfonylureas, meglitinides, insulin secretagogues, metformin, or α-glucosidase inhibitors) given as monotherapy, for at least 3 months prior to screening, and could discontinue that antihyperglycemic medication at Visit 2 (Week -2) and for the duration of the study. OR
* Untreated and had not taken any antihyperglycemic agent during the 2 months prior to screening; if not treated with an oral antihyperglycemic agent, the participant was considered by the investigator to have failed diet and exercise modification as the sole treatment for type 2 diabetes mellitus.
* Clinically stable in regard to medical conditions other than type 2 diabetes mellitus.
* Concomitant medications (other than oral antihyperglycemic agents) were at stable doses for at least 30 days prior to enrollment and were not anticipated to need adjustment during the study period.

Exclusion Criteria:

* History of type 1 diabetes and/or history of ketoacidosis.
* History of long-term (>2 months) therapy with insulin.
* History of prior treatment failure with, or intolerance of, a thiazolidinedione (ie, rosiglitazone, troglitazone, or pioglitazone).
* Treatment with a fibrate lipid-lowering agent (eg, fenofibrate, gemfibrozil).
* Confirmed repeat fasting glucose (≥2 readings of fasting blood glucose) >240 mg/dL (13.3 mmol/L) during the 2-week washout/stabilization and placebo run-in period (Period A).
* Body mass index (BMI) >45 kg/m2 at screening.
* History of weight loss >10% over the 3 months prior to screening.
* Female participant who was pregnant or breastfeeding.
* Systolic blood pressure ≥180 mmHg and/or diastolic blood pressure

  ≥110 mmHg.
* Any known history of congestive heart failure prior to screening.
* History of unstable angina, myocardial infarction, cerebrovascular accident, transient ischemic attack, or any revascularization within 6 months prior to screening. History of malignancy (except participants who had been disease-free for >10 years), or whose malignancy was a basal or squamous cell skin carcinoma. Any history of bladder cancer was an exclusion from participation. Women with a history of cervical dysplasia (CIN2 or higher) were to be excluded unless 2 consecutive normal cervical smears had subsequently been recorded prior to enrollment.
* Impaired liver function including evidence of acute or chronic hepatitis or liver disease by medical history, clinical signs or symptoms, or laboratory results.
* Evidence for ongoing infectious liver disease with positive hepatitis A antigen or immunoglobulin M antibody, hepatitis B surface antigen, or antibodies to hepatitis C virus. Participants with normal liver function tests and isolated positive antibodies to hepatitis B virus could have been included.
* Known (or evidence of) infection with human immunodeficiency virus.
* Known hemoglobinopathy or chronic anemia that required specific treatment within 5 years of the screening visit.
* History of alcohol or drug abuse within 1 year prior to screening.
* History of unstable major psychiatric disorders. Known or suspected allergy or hypersensitivity to thiazolidinedione agents.
* Clinically significant abnormalities in any pre-randomization laboratory analyses that, in the investigator's opinion, comprised an undue risk with the participant's participation, or could potentially confound results of the study.

Unexplained hematuria (>3 red blood cells per high-powered field by urine microscopy).

* Blood donation of ≥1 pint (0.5 liter) within the past 30 days prior to screening or plasma donation within 7 days prior to the screening visit (Visit 1).
* Prior known or possible exposure to rivoglitazone.
* Contraindication to treatment with pioglitazone once daily.
* Known or suspected allergy, hypersensitivity, or intolerance to the excipients of the investigational study medication.
* Participation in an interventional medical, surgical, or pharmaceutical study within 30 days prior to the screening visit (Visit 1).
* Any condition or concomitant therapy that, in the opinion of the investigator, might have posed a risk to the participant or made participation not in the participant's best interest.
* A direct or familial relationship with the Sponsor, investigator, or site personnel affiliated with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-11-14 (Actual); Primary Completion 2008-05-23 (Actual); Study Completion 2008-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (17):
- United States (17):
  - Huntsville, Alabama
  - San Diego, California
  - San Francisco, California
  - Ridgefield, Connecticut
  - Fort Lauderdale, Florida
  - Pembroke Pines, Florida
  - Port Gibson, Mississippi
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Kettering, Ohio
  - Fleetwood, Pennsylvania
  - Harrisburg, Pennsylvania
  - Simpsonville, South Carolina
  - Daingerfield, Texas
  - Dallas, Texas
  - Plano, Texas
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 94 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 73 clinic sites in the United States of America and 22 in India.
Pre-assignment Details: Participants with type 2 diabetes mellitus who were either untreated (ie, not receiving antihyperglycemic medication within at least 2 months prior to screening) or were treated with a single, non-thiazolidinedione agent as monotherapy without adequate glycemic control were enrolled in this study.
Groups:
- Placebo: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone-matching placebo tablet or a Pioglitazone-matching placebo capsule once daily for 18 weeks.
- Rivoglitazone 0.5mg: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone 0.5mg tablet once daily for 18 weeks.
- Rivoglitazone 1.0mg: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone 1.0mg tablet once daily for 18 weeks.
- Rivoglitazone 1.5mg: Participants with type 2 diabetes mellitus who were administered a Rivoglitazone 1.5mg tablet once daily for 18 weeks.
- Pioglitazone 15 mg: Participants with type 2 diabetes mellitus who were administered a Pioglitazone 15 mg capsule once daily for 18 weeks.
- Pioglitazone 30 mg: Participants with type 2 diabetes mellitus who were administered a Pioglitazone 30 mg capsule once daily for 18 weeks.
- Pioglitazone 45 mg: Participants with type 2 diabetes mellitus who were administered a Pioglitazone 45 mg capsule once daily for 18 weeks.
Period: Overall Study
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Started | 3 | 9 | 12 | 27 | 9 | 10 | 24
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 9 | 12 | 27 | 9 | 10 | 24
Not completed — Subject withdrew consent | 0 | 1 | 0 | 2 | 1 | 1 | 2
Not completed — Hyperglycemia meeting discontinuation criteria | 1 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Therapeutic failure/lack of efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Termination of study by Sponsor | 2 | 7 | 10 | 24 | 8 | 9 | 22
Not completed — Per medical monitor regarding thyroid-stimulating hormone level | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed from the All Randomized Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg | Total
Number analyzed (Participants) | 3 | 9 | 12 | 27 | 9 | 10 | 24 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (11.36) | 55.1 (13.03) | 58.3 (10.86) | 59.4 (10.46) | 57.0 (9.85) | 58.5 (7.71) | 58.0 (11.72) | 58.1 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 5 | 16 | 4 | 6 | 9 | 43
  Male | 2 | 7 | 7 | 11 | 5 | 4 | 15 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 4 | 3 | 2 | 4 | 2 | 18
  Not Hispanic or Latino | 3 | 6 | 8 | 24 | 7 | 6 | 22 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 3 | 1 | 0 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 6 | 0 | 2 | 8 | 20
  White | 1 | 8 | 9 | 18 | 8 | 7 | 12 | 63
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in A1c From Baseline Through Week 20 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Glycosylated hemoglobin (A1c) levels and mean changes in A1c were used to measure glycemic control. A1c categorical targets are <7.0% and <6.5%.
Time Frame: Baseline up to week 2, week 4, week 6, week 8, week 10, week 12, week 16, and week 20 post-dose.
Population: Change in A1c was assessed using the Full Analysis Set. There were "0" numbers analyzed reported beyond Week 6 due to early termination by the sponsor because of changes in the clinical development plan. Data was not collected for participants that did not complete the later time points prior to study termination so cannot be included in the table.
Measure: Mean (Standard Deviation); unit: percentage of A1c
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 3 | 9 | 12 | 27 | 8 | 10 | 24
percentage of A1c
  Baseline | 7.8 (0.55) | 7.5 (0.41) | 7.7 (0.67) | 7.5 (0.46) | 7.7 (0.56) | 7.5 (0.51) | 7.6 (0.50)
  Week 2: number analyzed (Participants) | 3 | 8 | 11 | 23 | 8 | 10 | 23
  Week 2 | 8.2 (0.87) | 7.6 (0.54) | 7.9 (0.96) | 7.6 (0.49) | 7.6 (0.61) | 7.5 (0.43) | 7.7 (0.56)
  Change in Baseline to Week 2: number analyzed (Participants) | 3 | 8 | 11 | 23 | 8 | 10 | 23
  Change in Baseline to Week 2 | 0.3 (0.67) | 0.1 (0.23) | 0.1 (0.54) | 0.1 (0.30) | -0.1 (0.23) | 0.1 (0.19) | 0.1 (0.31)
  Week 4: number analyzed (Participants) | 2 | 7 | 8 | 21 | 8 | 9 | 20
  Week 4 | 7.8 (1.06) | 7.6 (0.86) | 7.4 (0.42) | 7.5 (0.56) | 7.6 (0.68) | 7.4 (0.56) | 7.6 (0.62)
  Change from Baseline to Week 4: number analyzed (Participants) | 2 | 7 | 8 | 21 | 8 | 9 | 20
  Change from Baseline to Week 4 | -0.1 (0.28) | 0.2 (0.49) | -0.1 (0.32) | -0.0 (0.43) | -0.0 (0.32) | -0.1 (0.27) | -0.0 (0.37)
  Week 6: number analyzed (Participants) | 1 | 5 | 6 | 12 | 6 | 5 | 17
  Week 6 | 8.6 (NA) — Not available as data was calculated for one participant. | 7.7 (0.99) | 7.4 (0.39) | 7.3 (0.55) | 7.4 (0.68) | 7.2 (0.65) | 7.5 (0.73)
  Change from Baseline to Week 6: number analyzed (Participants) | 1 | 5 | 6 | 12 | 6 | 5 | 17
  Change from Baseline to Week 6 | 0.2 (NA) — Not available as data was calculated for one participant. | 0.3 (0.61) | -0.2 (0.25) | -0.1 (0.41) | -0.2 (0.18) | -0.2 (0.46) | -0.2 (0.44)
  Week 8: number analyzed (Participants) | 0 | 5 | 4 | 7 | 6 | 5 | 12
  Week 8 |  | 7.2 (0.62) | 7.4 (0.23) | 7.2 (0.52) | 7.6 (0.76) | 7.2 (0.54) | 7.4 (0.73)
  Change from Baseline to Week 8: number analyzed (Participants) | 0 | 5 | 4 | 7 | 6 | 5 | 12
  Change from Baseline to Week 8 |  | 0.0 (0.48) | -0.5 (0.53) | -0.2 (0.37) | 0.0 (0.78) | -0.2 (0.42) | -0.3 (0.47)
  Week 10: number analyzed (Participants) | 0 | 2 | 2 | 6 | 7 | 5 | 10
  Week 10 |  | 7.2 (0.92) | 7.2 (0.00) | 7.2 (0.40) | 7.6 (0.71) | 6.8 (0.70) | 7.2 (0.93)
  Change from Baseline to Week 10: number analyzed (Participants) | 0 | 2 | 2 | 6 | 7 | 5 | 10
  Change from Baseline to Week 10 |  | 0.0 (1.13) | -0.7 (0.28) | -0.3 (0.37) | -0.2 (0.27) | -0.4 (0.76) | -0.3 (0.58)
  Week 12: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
  Week 12 |  | 7.7 (NA) — Not available as data was calculated for one participant. | 7.2 (NA) — Not available as data was calculated for one participant. | 7.0 (0.54) | 7.2 (0.44) | 7.0 (0.39) | 7.0 (0.92)
  Change from Baseline to Week 12: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
  Change from Baseline to Week 12 |  | 0.7 (NA) — Not available as data was calculated for one participant. | -0.9 (NA) — Not available as data was calculated for one participant. | -0.2 (0.29) | -0.2 (0.29) | -0.1 (0.44) | -0.8 (0.50)
  Week 16: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 3
  Week 16 |  | 7.7 (NA) — Not available as data was calculated for one participant. |  |  |  | 6.9 (0.00) | 7.4 (0.60)
  Change from Baseline to Week 16: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 3
  Change from Baseline to Week 16 |  | 0.7 (NA) — Not available as data was calculated for one participant. |  |  |  | -0.4 (0.35) | -0.8 (0.67)
  Week 20: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Week 20 |  |  |  |  |  | 7.0 (NA) — Not available as data was calculated for one participant. | 7.4 (0.49)
  Change from Baseline to Week 20: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Change from Baseline to Week 20 |  |  |  |  |  | -0.6 (NA) — Not available as data was calculated for one participant. | -0.6 (0.42)

2. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline Through Week 20 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Normal fasting plasma glucose (FPG) -- or blood sugar -- is between 70 and 100 milligrams per deciliter (mg/dL) for people who do not have diabetes. People with Type 2 diabetes typically have FPG that is too high, so a negative change from baseline and a lower FPG means improvement.
Time Frame: Baseline up to week 2, week 4, week 6, week 8, week 12, week 16, and week 20 post-dose.
Population: Fasting Plasma Glucose was assessed from the Full Analysis Set. There were "0" numbers analyzed reported beyond Week 6 due to early termination by the sponsor because of changes in the clinical development plan. Data was not collected for participants that did not complete the later time points prior to study termination so cannot be included in the table.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 3 | 9 | 12 | 27 | 8 | 10 | 24
mg/dL
  Baseline | 218.7 (48.09) | 164.1 (45.09) | 160.1 (34.34) | 162.2 (42.37) | 173.3 (35.77) | 138.3 (22.89) | 158.5 (35.45)
  Week 2: number analyzed (Participants) | 3 | 8 | 11 | 22 | 8 | 10 | 24
  Week 2 | 210.0 (71.51) | 157.8 (48.45) | 149.8 (49.38) | 152.4 (50.06) | 160.8 (21.12) | 140.9 (19.43) | 144.7 (34.46)
  Change from Baseline to Week 2: number analyzed (Participants) | 3 | 8 | 11 | 22 | 8 | 10 | 24
  Change from Baseline to Week 2 | -8.7 (41.59) | -1.0 (20.06) | -10.5 (36.05) | -13.6 (33.75) | -12.5 (22.48) | 2.6 (16.93) | -13.8 (24.11)
  Week 4: number analyzed (Participants) | 2 | 7 | 8 | 21 | 8 | 9 | 20
  Week 4 | 157.5 (37.48) | 149.4 (55.44) | 128.6 (33.31) | 145.6 (35.32) | 171.4 (48.23) | 140.3 (30.49) | 143.6 (26.40)
  Change from Baseline to Week 4: number analyzed (Participants) | 2 | 7 | 8 | 21 | 8 | 9 | 20
  Change from Baseline to Week 4 | -33.5 (43.13) | -8.3 (12.50) | -24.6 (30.97) | -26.2 (27.69) | -1.9 (38.79) | 2.3 (20.34) | -20.0 (24.20)
  Week 6: number analyzed (Participants) | 1 | 5 | 6 | 12 | 7 | 5 | 16
  Week 6 | 218.0 (NA) — Not available as data was calculated for one participant. | 158.4 (54.77) | 126.5 (24.14) | 126.9 (17.76) | 174.3 (41.80) | 134.0 (25.00) | 146.8 (44.22)
  Change from Baseline to Week 6: number analyzed (Participants) | 1 | 5 | 6 | 12 | 7 | 5 | 16
  Change from Baseline to Week 6 | 31.0 (NA) — Not available as data was calculated for one participant. | -0.2 (23.70) | -30.8 (22.22) | -41.1 (33.09) | 0.7 (48.65) | -4.0 (12.51) | -17.1 (41.99)
  Week 8: number analyzed (Participants) | 0 | 5 | 4 | 7 | 6 | 5 | 12
  Week 8 |  | 153.6 (56.44) | 129.5 (15.35) | 125.0 (15.70) | 149.2 (35.72) | 145.6 (49.47) | 148.3 (34.55)
  Change from Baseline to Week 8: number analyzed (Participants) | 0 | 5 | 4 | 7 | 6 | 5 | 12
  Change from Baseline to Week 8 |  | 12.2 (32.89) | -41.3 (26.29) | -35.1 (20.51) | -23.2 (57.14) | 7.6 (41.71) | -20.0 (28.27)
  Week 12: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
  Week 12 |  | 142.0 (NA) — Not available as data was calculated for one participant. | 131.0 (NA) — Not available as data was calculated for one participant. | 120.3 (11.79) | 131.7 (13.43) | 122.3 (13.23) | 126.4 (27.77)
  Change from Baseline to Week 12: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
  Change from Baseline to Week 12 |  | 16.0 (NA) — Not available as data was calculated for one participant. | -51.0 (NA) — Not available as data was calculated for one participant. | -32.5 (25.38) | -25.3 (18.58) | -9.8 (25.08) | -29.4 (20.50)
  Week 16: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 3
  Week 16 |  | 159.0 (NA) — Not available as data was calculated for one participant. |  |  |  | 111.0 (2.83) | 133.7 (22.19)
  Change from Baseline to Week 16: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 2 | 3
  Change from Baseline to Week 16 |  | 33.0 (NA) — Not available as data was calculated for one participant. |  |  |  | -19.5 (4.95) | -39.3 (51.78)
  Week 20: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Week 20 |  |  |  |  |  | 107.0 (NA) — Not available as data was calculated for one participant. | 124.0 (15.56)
  Change from Baseline to Week 20: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Change from Baseline to Week 20 |  |  |  |  |  | -25.0 (NA) — Not available as data was calculated for one participant. | -18.0 (1.41)

3. Secondary Outcome: Change in Total Cholesterol From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Total cholesterol is a measure of the total amount of cholesterol in the blood, including low-density lipoprotein cholesterol (LDL-C) - the "bad" cholesterol, high-density lipoprotein cholesterol (HDL-C) - the "good" cholesterol, and triglycerides. The equation to calculate total cholesterol is: LDL + HDL + (triglycerides/5) = total cholesterol.
Time Frame: Baseline up to week 12 post-dose.
Population: Total cholesterol was assessed from the Full Analysis Set. There were "0" numbers analyzed reported beyond Week 6 due to early termination by the sponsor because of changes in the clinical development plan. Data was not collected for participants that did not complete the later time points prior to study termination so cannot be included in the table.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 3 | 9 | 12 | 27 | 8 | 10 | 24
mg/dL
  Baseline | 162.2 (38.10) | 211.3 (52.87) | 204.9 (63.66) | 171.6 (38.95) | 172.1 (35.49) | 201.7 (50.13) | 188.1 (47.45)
  Week 12: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
  Week 12 |  | 311.0 (NA) — Not available as data was calculated for one participant. | 193.0 (NA) — Not available as data was calculated for one participant. | 145.8 (17.27) | 151.3 (47.08) | 213.3 (28.62) | 186.6 (36.19)

4. Secondary Outcome: Percent Change in Total Cholesterol From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: as for outcome 3
Time Frame: Baseline up to week 12 post-dose.
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
percent change |  | 8.9 (NA) — Not available as data was calculated for one participant. | -8.5 (NA) — Not available as data was calculated for one participant. | -2.2 (6.46) | -1.6 (9.54) | 2.7 (15.73) | 7.4 (15.60)

5. Secondary Outcome: Change in Total Triglycerides From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Total Triglycerides (TG) is a measure of the total amount of triglycerides in the blood. The equation to calculate total triglycerides is: (total cholesterol-Low-density Lipoprotein cholesterol (LDL- C) - High-density lipoprotein cholesterol (HDL- C)) x 5 = Total Triglycerides. A negative change means improvement.
Time Frame: Baseline up to week 12 post-dose.
Population: Total Triglycerides were assessed from the Full Analysis Set. There were "0" numbers analyzed reported beyond Week 6 due to early termination by the sponsor because of changes in the clinical development plan. Data was not collected for participants that did not complete the later time points prior to study termination so cannot be included in the table.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 3 | 9 | 12 | 27 | 8 | 10 | 24
mg/dL
  Baseline | 100.8 (15.94) | 293.2 (300.50) | 214.8 (145.63) | 156.5 (85.96) | 165.7 (118.31) | 221.0 (188.82) | 163.0 (72.29)
  Week 12: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
  Week 12 |  | 179.0 (NA) — Not available as data was calculated for one participant. | 180.0 (NA) — Not available as data was calculated for one participant. | 72.0 (6.73) | 82.3 (44.52) | 161.3 (100.69) | 90.8 (41.95)

6. Secondary Outcome: Percent Change in Total Triglycerides From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: as for outcome 5
Time Frame: Baseline up to week 12 post-dose.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
percent change |  | -15.4 (NA) — Not available as data was calculated for one participant. | -34.1 (NA) — Not available as data was calculated for one participant. | -16.8 (16.17) | -20.5 (40.04) | -16.1 (24.80) | -16.2 (33.60)

7. Secondary Outcome: Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Low-density lipoprotein cholesterol (LDL-C) is a measure of the total amount of low-density lipoprotein cholesterol in the blood. LDL-C was measured as part of the fasting lipid panel. LDL-C is considered "bad" cholesterol, so a lower score (negative change) means improvement.
Time Frame: Baseline up to week 12 post-dose.
Population: Low-Density Lipoprotein Cholesterol was assessed from the Full Analysis Set. There were "0" numbers analyzed reported beyond Week 6 due to early termination by the sponsor because of changes in the clinical development plan. Data was not collected for participants that did not complete the later time points prior to study termination so cannot be included in the table.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 3 | 9 | 12 | 27 | 8 | 10 | 24
mg/dL
  Baseline: number analyzed (Participants) | 3 | 8 | 11 | 27 | 8 | 9 | 24
  Baseline | 101.7 (33.90) | 124.1 (45.67) | 125.8 (53.79) | 95.9 (28.52) | 95.7 (22.73) | 105.8 (35.12) | 108.4 (41.93)
  Week 12: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
  Week 12 |  | 226.0 (NA) — Not available as data was calculated for one participant. | 112.0 (NA) — Not available as data was calculated for one participant. | 78.5 (20.70) | 82.7 (45.54) | 129.8 (10.56) | 111.6 (24.67)

8. Secondary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: as for outcome 7
Time Frame: Baseline up to week 12 post-dose.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 3 | 5
percent change |  | 16.8 (NA) — Not available as data was calculated for one participant. | -1.8 (NA) — Not available as data was calculated for one participant. | -8.6 (3.25) | -5.7 (18.70) | 14.5 (1.15) | 14.0 (18.48)

9. Secondary Outcome: Change in High-Density Lipoprotein Cholesterol From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: High-density lipoprotein cholesterol (HDL-C) is a measure of the total amount of high-density lipoprotein cholesterol in the blood. HDL-C was measured as part of the fasting lipid panel. HDL-C is considered "good" cholesterol, so a higher score (positive change) means improvement.
Time Frame: Baseline up to week 12 post-dose.
Population: High-Density Lipoprotein Cholesterol was assessed from the Full Analysis Set. There were "0" numbers analyzed reported beyond Week 6 due to early termination by the sponsor because of changes in the clinical development plan. Data was not collected for participants that did not complete the later time points prior to study termination so cannot be included in the table.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 3 | 9 | 12 | 27 | 8 | 10 | 24
mg/dL
  Baseline | 40.2 (2.31) | 43.9 (10.84) | 42.4 (9.23) | 44.3 (13.70) | 42.5 (10.87) | 49.4 (14.23) | 47.2 (11.86)
  Week 12: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
  Week 12 |  | 49.0 (NA) — Not available as data was calculated for one participant. | 45.0 (NA) — Not available as data was calculated for one participant. | 52.8 (11.53) | 52.3 (21.01) | 51.3 (10.14) | 56.6 (14.43)
  Change from Baseline Week 12: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
  Change from Baseline Week 12 |  | -1.0 (NA) — Not available as data was calculated for one participant. | 5.9 (NA) — Not available as data was calculated for one participant. | 13.1 (14.03) | 12.9 (12.93) | 10.8 (10.26) | 11.1 (10.39)

10. Secondary Outcome: Percent Change in High-Density Lipoprotein Cholesterol From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: as for outcome 9
Time Frame: Baseline up to week 12 post-dose.
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
percent change |  | -1.0 (NA) — Not available as data was calculated for one participant. | 5.9 (NA) — Not available as data was calculated for one participant. | 13.1 (14.03) | 12.9 (12.93) | 10.8 (10.26) | 11.1 (10.39)

11. Secondary Outcome: Change in Apolipoprotein (Apo) A-I From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Apolipoprotein (Apo) A-I is a measure of the total amount of Apolipoprotein (Apo) A-I in the blood. Apo A-I was measured as part of the fasting lipid panel.
Time Frame: Baseline up to week 12 post-dose.
Population: Apolipoprotein (Apo) A-I was assessed from the Full Analysis Set. There were instances of zero (0) numbers analyzed reported beyond Week 6 due to early termination by the sponsor because of changes in the clinical development plan. Data was not collected for participants that did not complete the later time points prior to study termination and were not reported in the table.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 3 | 9 | 12 | 27 | 8 | 10 | 24
mg/dL
  Baseline | 134.0 (7.57) | 146.7 (15.68) | 139.7 (16.20) | 142.4 (27.72) | 133.0 (20.34) | 158.6 (31.57) | 149.6 (25.89)
  Week 12: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
  Week 12 |  | 144.0 (NA) — Not available as data was calculated for one participant. | 141.0 (NA) — Not available as data was calculated for one participant. | 149.8 (21.08) | 145.3 (34.27) | 153.0 (24.14) | 158.2 (31.44)

12. Secondary Outcome: Percent Change in Apolipoprotein (Apo) A-I From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: as for outcome 11
Time Frame: Baseline up to week 12 post-dose.
Population: Apolipoprotein (Apo) A-I was assessed from the Full Analysis Set. There were instances of zero (0) number analyzed reported beyond Week 6 due to early termination by the sponsor because of changes in the clinical development plan. Data were not collected for participants that did not complete the later time points prior to study termination and not available for the table.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
percent change |  | -14.5 (NA) — Not available as data was calculated for one participant. | -2.8 (NA) — Not available as data was calculated for one participant. | 2.8 (9.18) | 3.0 (6.90) | 0.3 (6.81) | 1.4 (10.19)

13. Secondary Outcome: Change in Apolipoprotein (Apo) B From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Apolipoprotein (Apo) B is a measure of the total amount of Apolipoprotein (Apo) B in the blood. Apo B was measured as part of the fasting lipid panel.
Time Frame: Baseline up to week 12 post-dose.
Population: Apolipoprotein (Apo) B was assessed from the Full Analysis Set. There were instances of zero (0) number analyzed reported beyond Week 6 due to early termination by the sponsor because of changes in the clinical development plan. Data were not collected for participants that did not complete the later time points prior to study termination and not available for the table.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 3 | 9 | 12 | 27 | 8 | 10 | 24
mg/dL
  Baseline | 94.0 (26.44) | 119.1 (36.53) | 121.9 (36.37) | 101.3 (29.72) | 105.5 (34.32) | 113.4 (25.20) | 108.4 (31.94)
  Week 12: number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
  Week 12 |  | 206.0 (NA) — Not available as data was calculated for one participant. | 115.0 (NA) — Not available as data was calculated for one participant. | 76.5 (17.06) | 77.7 (31.53) | 120.8 (15.46) | 95.6 (23.39)

14. Secondary Outcome: Percent Change in Apolipoprotein (Apo) B From Baseline Through Week 12 Following Rivoglitazone Compared to Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: as for outcome 13
Time Frame: Baseline up to week 12 post-dose.
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 0 | 1 | 1 | 4 | 3 | 4 | 5
percent change |  | 13.2 (NA) — Not available as data was calculated for one participant. | -12.2 (NA) — Not available as data was calculated for one participant. | -11.5 (5.21) | -14.8 (20.97) | 0.1 (6.63) | 1.7 (16.20)

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events by System Organ Class and Preferred Term Following Rivoglitazone or Pioglitazone as Monotherapy Treatment of Type 2 Diabetes Mellitus
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that occurred on or after the first dose of randomized study medication and ongoing adverse events that started prior to the first dose of randomized study medication and increased in severity on or after the first dose of randomized study medication.
Time Frame: Baseline up to week 26 post-dose, approximately a total of 27 weeks.
Population: Treatment-emergent adverse events were assessed from the Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
Number analyzed (Participants) | 3 | 9 | 12 | 27 | 8 | 10 | 24
Participants
  Lymphadenitis | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypothyroidism | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Conjunctivitis | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Eye Pruritus | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Ocular Hyperaemia | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Abdominal Pain | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Dry Mouth | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Flatulence | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Stomach Discomfort | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Malaise | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Non-cardiac chest pain | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Oedema | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Oedema peripheral | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Cholelithiasis | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Seasonal allergy | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Bronchitis | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Fungal infection | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Furuncle | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Influenza | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Nasopharyngitis | 0 | 0 | 1 | 1 | 0 | 0 | 1
  Sinusitis | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Upper respiratory tract | 0 | 0 | 0 | 2 | 1 | 1 | 1
  Viral upper respiratory tract infection | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Arthropod bite | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Back injury | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Haemoglobin decreased | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Red blood cell morphology abnormal | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Back pain | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Flank pain | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Joint crepitation | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Muscle twitching | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Musculoskeletal pain | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Musculoskeletal stiffness | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Myalgia | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Pain in extremity | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Carpal tunnel syndrome | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Dizziness | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Headache | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Insomnia | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Mood altered | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Pharyngolaryngeal pain | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperhidrosis | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Rash | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypertension | 0 | 1 | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event (TEAE) data were collected from Baseline (Day 1) up to week 26 post-dose, approximately a total of 27 weeks.
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events (AEs) that occurred on or after the first dose of randomized study medication and ongoing adverse events that started prior to the first dose of randomized study medication and increased in severity on or after the first dose of randomized study medication.
Arm/Group | Placebo | Rivoglitazone 0.5mg | Rivoglitazone 1.0mg | Rivoglitazone 1.5mg | Pioglitazone 15 mg | Pioglitazone 30 mg | Pioglitazone 45 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/9 | 0/12 | 0/27 | 0/8 | 0/10 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/9 | 0/12 | 0/27 | 0/8 | 0/10 | 0/24
Other Adverse Events (participants affected / at risk) | 0/3 | 5/9 | 1/12 | 8/27 | 4/8 | 2/10 | 10/24
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3) | Rivoglitazone 0.5mg (N=9) | Rivoglitazone 1.0mg (N=12) | Rivoglitazone 1.5mg (N=27) | Pioglitazone 15 mg (N=8) | Pioglitazone 30 mg (N=10) | Pioglitazone 45 mg (N=24)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Edema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Edema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Red blood cell morphology abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No